CLINICAL TRIAL: NCT02149225
Title: A Phase I Trial of Actively Personalized Peptide Vaccinations Plus Immunomodulators in Patients With Newly Diagnosed Glioblastoma Concurrent to First Line Temozolomide Maintenance Therapy
Brief Title: GAPVAC Phase I Trial in Newly Diagnosed Glioblastoma Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Immatics Biotechnologies GmbH (Industry)
Collaborators: BioNTech SE (Industry); University Hospital Tuebingen (Other); BCN Peptides (Industry); EU-funded GAPVAC Consortium (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GAPVAC-101; 2013-002801-71 (EudraCT Number)
Record Dates: First submitted 2014-05-16; First posted 2014-05-29 (Estimated); Last update posted 2018-08-07 (Actual); Status verified 2018-08

CONDITIONS: Glioblastoma
Keywords: Actively personalized peptide vaccinations; Newly diagnosed Glioblastoma; Concurrent to first line temozolomide maintenance therapy
MeSH Terms: conditions — Glioblastoma | interventions — poly ICLC; Granulocyte-Macrophage Colony-Stimulating Factor; sargramostim

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- APVAC1 and 2 vaccine plus polyICLC and GMCSF concurrent to TMZ (Experimental)
  Interventions: Drug: APVAC1 vaccine plus Poly-ICLC and GM-CSF; Drug: APVAC2 vaccine plus Poly-ICLC and GM-CSF

INTERVENTIONS:
Drug: APVAC1 vaccine plus Poly-ICLC and GM-CSF — APVAC1 vaccines (i.d.) will be individually assembled for each patient and can be applied to the patient approx. 3 months after enrollment. APVAC1 drug products are composed of 5 to 10 peptides from the GAPVAC warehouse. The APVAC1 vaccine will be applied concurrent to maintenance TMZ cycles after completion of chemoradiation therapy (CRT). Beginning on day 15 of the first maintenance TMZ cycle, patients will receive 11 vaccinations with APVAC1 drug products during 22 weeks. 578 μg per peptide per vial are used.
  Poly ICLC (1.5 mg s.c.) will be used as immunomodulator with all vaccinations except the second applications of APVAC1 (Day 2) and APVAC2 vaccines (Day 2*) to avoid dose accumulation on consecutive days.
  The 2. immunomodulator GM-CSF (75 μg) will be applied i.d. with the first six vaccinations with both vaccines, APVAC1 and APVAC2. A total of 12 GM-CSF doses will be applied. GM-CSF will be applied to the APVAC vaccination site 10-30 min before injection of the APVACs.
  Other Names: Actively Personalized Vaccine; Hiltonol; Leukine
Drug: APVAC2 vaccine plus Poly-ICLC and GM-CSF — APVAC2 vaccines (i.d.) will be ready for use ca. 6 months after enrollment, as these peptides have to be newly synthesized for each patient following identification of the mutanome and corresponding mutated peptides in the HLA ligandome. APVAC2 drug products are composed of 1 or 2 peptides de novo synthesized for an individual patient. Patients will be repeatedly vaccinated with APVAC2 drug products beginning on day 15 of the 4. maintenance TMZ cycle. Patients will receive 8 vaccinations within 10 weeks. 578 μg per peptide per vial are used.
  Poly-ICLC (1.5 mg s.c.) will be used as immunomodulator with all vaccinations except the second applications of APVAC1 (Day 2) and APVAC2 vaccines (Day 2*) to avoid dose accumulation on consecutive days.
  GM-CSF (75 μg) will be applied i.d. with the first six vaccinations with both vaccines, APVAC1 and APVAC2. A total of 12 GM-CSF doses will be applied. GM-CSF will be applied to the APVAC vaccination site 10-30 min before injection of the APVACs.
  Other Names: Actively Personalized Vaccine; Hiltonol; Leukine

SUMMARY:
The primary objective of this study is to assess the safety and tolerability, feasibility and biological activity (immunogenicity) of the actively personalized vaccination (APVAC) concept in newly diagnosed glioblastoma (GB) patients.

DETAILED DESCRIPTION:
This is a multicenter, open-label, single arm, first-in-man phase I trial to investigate the safety, feasibility and immunogenicity of the novel APVAC approach in patients with newly diagnosed GB.

Primary Endpoints:

* Safety: Determine the safety and tolerability profile of patient-tailored APVAC vaccines when administered with immunomodulators concurrent to maintenance temozolomide (TMZ) cycles.
* Feasibility: Determine duration and success rates for APVAC1 and APVAC2 processes and for vaccinations with APVAC drug products.
* Biological activity: Descriptive analysis of induced T-cell responses after vaccinations with APVAC1 and APVAC2 drug products plus immunomodulators.

Secondary Study Objectives:

* Identification of biomarkers putatively predictive for immunological response and/or associated with clinical success or failure. Analyzed biomarkers may include non-cellular parameters measured from tumor, plasma or serum, and cellular parameters measured from peripheral blood mononuclear cells (PBMCs), leukapheresis samples or isolated tumor-infiltrating lymphocytes (TILs).
* Description of potential clinical activity of the APVAC drug products. Descriptive analysis of clinical outcome in patients will be reported including OS and PFS. Correlation analysis of these parameters with immune response data may provide first hints on clinical activity of the vaccine.

After the standard chemoradiotherapy with TMZ has been completed and as soon as the start of the first maintenance TMZ cycle the vaccination phase begins. It starts with the first APVAC1 vaccination, followed by additional APVAC2 vaccinations at a later time point and ends with the Last Endpoint Evaluation Visit (LEEV) of a patient.

Single vaccinations with APVAC vaccines consist of an intradermal (i.d.) injection of the personalized APVAC drug product into the skin of the thigh, shoulder or abdomen followed by subcutaneous (s.c.) injection of 1.5 mg poly-ICLC (Hiltonol®) in close proximity to the vaccination site. The second immunomodulator GM-CSF (75 μg) will be applied i.d. to the APVAC vaccination site 10-30 min before injection of the APVACs.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed, newly diagnosed GB (astrocytoma WHO grade IV)
2. HLA phenotype defined by warehouse composition (HLA-A*02:01 or HLA-A*24:02 positive patients only; both as determined by a PCR-based 4-digit typing method)
3. Gross total resection (as defined by less than 1 cm2 residual tumor mass on the largest perpendicular axes in post-operative scan taken within 48 h post-surgery; standard MRI conformable to the present national and international guidelines is sufficient)
4. At least 0.5 g tumor tissue freshly cryopreserved during surgery
5. Age ≥18 years
6. KPS ≥70%
7. Life expectancy > 6 months
8. Patient is a candidate for and willing to receive standard CRT with TMZ followed by maintenance TMZ cycles
9. Patient is not on steroids or on stable or decreasing steroid levels not exceeding 2 mg/day dexamethasone (or equivalent doses of other steroids) during the last 3 days prior to enrollment
10. Absolute lymphocyte count (ALC) >1.0 x109/L (re-screening of lymphocyte counts is allowed)
11. Ability of subject to understand and the willingness to sign written informed consent for study participation. Written consent by a legally authorized representative is not sufficient.
12. Availability of an APVAC analysis and manufacturing slot confirmed by the sponsor
13. Female patients who are post-menopausal (no menstrual period for a minimum of 1 year), or surgically sterile (bilateral tubal ligation, bilateral oophorectomy, or hysterectomy), practice one of the following medically acceptable methods of birth control (hormonal methods, intrauterine device or double-barrier methods) or practice total abstinence
14. Male patients willing to use contraception (condoms with spermicidal jellies or cream) upon study entry and during the course of the study, have undergone vasectomy or are practicing total abstinence

Exclusion Criteria:

1. Abnormal (≥ Grade 2 CTCAE v4.0) laboratory values for hematology, liver and renal function (serum creatinine). In detail the following values apply as exclusion criteria:

   1. Hemoglobin < 10 g/dL (6.2 mmol/L)
   2. White blood cell count (WBC) decrease (<3.0 x109/L) or increase (>10.0 x109/L)
   3. Absolute neutrophil count (ANC) decrease < 1.5 x109/L
   4. Platelet count decrease < 75 x109/L
   5. Bilirubin > 1.5 x ULN (upper limit of normal according to the performing lab's reference range)
   6. ALAT > 3 x ULN
   7. ASAT > 3 x ULN
   8. GGT6 > 2.5 x ULN
   9. Serum creatinine increased > 1.5 x ULN
2. HIV infection or active Hepatitis B or C infection, or active infections requiring oral or intravenous antibiotics or that can cause a severe disease and pose a severe danger to lab personnel working on patients' blood or tissue (e.g. rabies).
3. Prior therapy for glioma (except surgery and steroids) including but not limited to carmustine wafers and immunotherapy
4. Any condition contraindicating leukapheresis from peripheral veins
5. Concurrent participation in another interventional clinical trial studying a drug or treatment regimen.
6. Clinically relevant autoimmune diseases (with the exception of thyroid diseases)
7. Immunosuppression, not related to prior treatment for malignancy, or prior drug reaction
8. Any condition that in the judgment of the investigator interferes with the probability that an individual patient may receive and benefit from APVAC vaccinations (e.g. high risk of early disease progression / recurrence; immunocompromised status; anticipated compliance problems)
9. Serious illness or condition, which according to the investigator, poses an undue risk for the patient when participating in the trial, including, but not limited to, any of the following:

   * Clinically significant cardiovascular disease
   * New York Heart Association class III-IV congestive heart failure
   * Symptomatic peripheral vascular disease
   * Severe pulmonary dysfunction
   * Severe diabetes
   * Severe mental retardation
10. History of other malignancies (except for adequately treated basal or squamous cell carcinoma or carcinoma in situ) within the last 5 years unless the patient has been disease-free for 5 years
11. Pregnancy or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2014-10; Primary Completion 2018-06 (Actual); Study Completion 2018-06 (Actual)

PRIMARY OUTCOMES:
Safety profile of patient-tailored APVAC vaccines when administered with immunomodulators concurrent to maintenance TMZ cycles | Continously for about 40 weeks plus follow-up
  Number of Adverse Events (AEs) and Serious Adverse Events (SAEs) and percentage of patients with AEs and SAEs (listed per grade and MedDRA (Medical Dictionary for Regulatory Activities ) preferred terms) will be reported.
Frequency of CD8 T cells specific for vaccinated APVAC peptides as measure of immunological response to and biological activity of the vaccine | Till 17 weeks of vaccination
  To analyze whether vaccinations with APVAC drug products plus poly-ICLC and GM-CSF induce immune responses in the patients. Peripheral blood mononuclear cells will be analyzed for the presence and functionality of T cells recognizing the peptides vaccinated within the individualized APVACs.
  * Immunogenicity rate: Number of vaccine induced T-cell responses normalized to the number of peptides vaccinated.
  * Immune responder rate: Number of patients with at least one vaccine induced T-cell response
  * Multi-TUMAP responder rate: Number of patients with at least two vaccine induced T-cell response
  * Average number of immune responses per patient

SECONDARY OUTCOMES:
Frequency of immune cell populations in the blood and concentrations of a large panel of serum and plasma proteins with immunological relevance as a measure of the immune status of the patient | Up to 10 months
  Putatively predictive for immunological response and/or associated with clinical success or failure. Analyzed biomarkers may include non-cellular parameters measured from tumor, plasma or serum, and cellular parameters measured from peripheral blood mononuclear cells (PBMCs), leukapheresis samples or isolated tumor-infiltrating lymphocytes (TILs).
Overall survival | 2018 (estimated)
  Median OS, the survival rate at one and at two years will be reported
Progression-free survival | At 6 months
  Median progression free survival (PFS) and PFS rates at 6 months will be described for patients in the safety and per protocol populations

CONTACTS AND LOCATIONS:
Overall Officials: Wolfgang Wick, Professor, Principal Investigator — University of Heidelberg Medical Center; Pierre-Yves Dietrich, Professor, Principal Investigator — University Hospital, Geneva
Locations (6):
- Rigshospitalet, The Finsen Centre, Department of Oncology, Copenhagen, Denmark
- Germany (2):
  - Neurologische Klinik & Nationales Centrum für Tumorerkrankungen Heidelberg, Heidelberg
  - Zentrum für Neurologie und Klinik für Neurochirurgie, Tübingen
- Leiden University Medical Center, Department of Medical Oncology, Leiden, Netherlands
- Vall d'Hebron University Hospital, Barcelona, Spain
- Hôpitaux Universitaires de Genève, Geneva, Switzerland